CLINICAL TRIAL: NCT04009551
Title: Zekai Tahir Burak Women's Health Research and Education Hospital
Brief Title: Epidemiology, Treatment and Prognosis of Neonatal Meningitis in Turkey: A Multicenter Study
Acronym: NEO-MENINGITIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta Oncel, Head of Neonatology, Tepecik Training and Research Hospital
Other Study IDs: Tepecik35
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Neonatal Meningitis
Keywords: meningitis; epidemiology; neonate; newborn
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Meningitis, defined as inflammation of the meninges caused by different pathogens, is a serious infection associated with high morbidity and mortality. It occurs more commonly in the neonatal period than in any other age group. Neonatal meningitis is a devastating infection that occurs more commonly in neonates than in any other age group, and is associated with significant morbidity and mortality. In this study, we aimed to evaluate epidemiology, treatment and prognosis of neonatal meningitis in a large-scale retrospective multicenter cohort study.

The main objectives of this study were to assess the incidence, temporal trend, risk factors, causative organisms, and short term outcomes of neonatal meningitis in a large national cohort of newborn infants admitted to Turkey NICUs.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a positive cerebrospinal fluid culture/PCR of bacterial pathogen.
* Subject has a positive blood culture of bacterial pathogen and counts of white blood cells in cerebrospinal fluid ≥20 /mm3.

Exclusion Criteria:

* Major congenital anomalies
* Cultures positive for coagulase-negative staphylococci (CONS) were excluded as possible contaminants, if not clinically and laboratory compatible with meningitis.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In this study,
  1. Lumbar puncture performed due to suspected meningitis and
  2. CSF laboratory findings are consistent with meningitis and
  3. Positivity in CSF culture and/or CSF PCR
  4. Neonates hospitalized between 1 January 2014 and 31 May 2019 will be included in the study.
     * The list of all cases diagnosed as on Neonatal Meningitis with growth in CSF culture and / or causative agent by CSF PCR will be obtained from the hospital's database.
     * Term infants will be included in the study until 1 month and preterm infants will be adjusted until the first month.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of neonatal meningitis | average of 5 years
  Occurrence of a meningitis in NICU within a specified period of time. (Number of neonatal meningitis cases / Total number of inpatients in the study period)

SECONDARY OUTCOMES:
Causative organisms | average of 5 years
  Number and types of isolated microorganisms in CSF cultures
Neurodevelopmental Outcome | 18 to 24 months
  - Bayley Scales of Infant Development, Second Edition (BSID II), was performed a comprehensive assessment including neurological and developmental evaluation. The mean BSID II score is 100 for Mental Developmental Index (MDI) and Psychomotor Developmental Index (PDI), with a standard deviation (SD) of 15; a score of less than 70 (42 SDs below the mean) indicates a significant delay. Infants who were so severely impaired that testing with the BSID II could not be performed were assigned a MDI and PDI score of 49.
Mortality | up to 28 days
  Neonatal meningitis related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yekta Oncel, M.D., Principal Investigator — Tepecik Training and Research Hospital
Locations (5):
- Turkey (Türkiye) (5):
  - Zekai Tahir Burak Women's Health Research and Education Hospital, Ankara
  - Bursa Yuksek Ihtisas Research and Education Hospital, Bursa
  - Gazi Yasargil Education Research Hospital, Diyarbakır
  - İstanbul Kanuni Sultan Süleyman Training and Research Hospital, Istanbul
  - Izmir Katip Celebi University, Medical Faculty, Izmir

IPD SHARING:
Plan to Share IPD: Undecided